CLINICAL TRIAL: NCT02637024
Title: A Phase II Randomized Trial of Radiation Fractionation Schedules for Once-a-Day Accelerated Partial Breast Irradiation (OPAR)
Brief Title: Trial of Radiation Fractionation Schedules for Once-a-Day Accelerated Partial Breast Irradiation
Acronym: OPAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Canadian Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OCOG-2015-OPAR
Record Dates: First submitted 2015-12-16; First posted 2015-12-22 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer; DCIS
Keywords: Breast Cancer; DCIS; Radiotherapy; Partial breast irradiation; Radiation fractions
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- APBI: 30 Gy (Experimental): Radiotherapy of 3 Dimensional Conformal Radiation Therapy (3DCRT) Accelerated Partial Breast Irradiation (APBI) 30 Gy in 5 daily fractions of 6 Gy
  Interventions: Radiation: APBI: 30 Gy
- APBI: 27.5 Gy (Experimental): Radiotherapy of 3 Dimensional Conformal Radiation Therapy (3DCRT) Accelerated Partial Breast Irradiation (APBI) 27.5 Gy in 5 daily fractions of 5.5 Gy
  Interventions: Radiation: APBI: 27.5 Gy

INTERVENTIONS:
Radiation: APBI: 30 Gy — 30 Gy in 5 fractions of 6 Gy, delivered daily, Monday to Friday, over a period of 5-8 days. A multiple small field 3D-conformal or intensity modulated radiation therapy (IMRT) technique will be used.
  Arms: APBI: 30 Gy
Radiation: APBI: 27.5 Gy — 27.5 Gy in 5 fractions of 5.5 Gy, delivered daily, Monday to Friday, over a period of 5-8 days. A multiple small field 3D-conformal or intensity modulated radiation therapy (IMRT) technique will be used.
  Arms: APBI: 27.5 Gy

SUMMARY:
This is a multi-centre randomized phase II trial in women with invasive carcinoma of the breast with negative axillary nodes or Ductal Carcinoma In-situ (DCIS) treated by Breast Conserving Surgery (BCS). Eligible, consenting patients will be randomly allocated to receive radiotherapy of 3 Dimensional Conformal Radiation Therapy (3DCRT) Accelerated Partial Breast Irradiation (APBI) 30 Gray (Gy) in 5 daily fractions of 6Gy or 27.5Gy in 5 daily fractions of 5.5Gy over one week. Patients will be followed at 12, 24, 36 and 60 months post randomization. Cosmetic outcome will be measured using photographs and evaluated by a panel of trained radiation oncologists. Radiation toxicity will be assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE).

DETAILED DESCRIPTION:
Women with invasive carcinoma of the breast with negative axillary nodes or DCIS, following BCS and/or chemotherapy, who meet the inclusion criteria will be screened and approached for eligibility assessment and potential study enrollment. All potentially eligible and consenting patients who do not meet the exclusion criteria will have a Computed Tomography (CT) simulation of the ipsilateral breast prior to randomization. All cases will be required to be planned prior to the randomization to ensure that dosimetric coverage and normal tissue restrictions can be met. If the seroma is not clearly visible or if the surgical clips do not adequately identify a previous surgical cavity, the patient will not be eligible for randomization.

Eligible, consenting patients will be randomly allocated to receive radiotherapy of 3DCRT APBI 30Gy in 5 daily fractions of 6Gy or 27.5Gy in 5 daily fractions of 5.5Gy over one week. Patients will be followed at 12, 24, 36 and 60 months post randomization. Cosmetic outcome will be measured using photographs and evaluated by a panel of trained radiation oncologists using the EORTC Breast Cosmetic Rating System. Radiation toxicity will be assessed using the NCI CTCAE version 4.02. The primary outcome is adverse cosmetic outcome at 2 years. The trial will be conducted in clinical centres within Canada.

ELIGIBILITY:
Inclusion Criteria:

1. Females with a new histological diagnosis of DCIS or invasive carcinoma of the breast with no evidence of metastatic disease.
2. Treated by BCS with microscopically clear resection margins for invasive and non-invasive disease (or no residual disease on re-excision).
3. Negative axillary node involvement, including positive cells only identified by Immunohistochemistry (IHC) as determined either by sentinel node biopsy or axillary node dissection, or a clinical exam for patients with DCIS only.

Exclusion Criteria:

1. Age less than 50 years
2. Known to be Breast Cancer Type 1 Susceptibility Protein (BRCA 1) and/or Breast Cancer Type 2 Susceptibility Protein (BRCA 2) positive
3. Tumour size >3 cm in greatest diameter on pathological examination (including the invasive and non-invasive components)
4. Tumour invades the skin (i.e. T4 disease)
5. Tumour histology limited to lobular carcinoma only
6. Grade III invasive breast carcinoma or nuclear grade III for patients with DCIS alone
7. Triple negative invasive breast cancer
8. Her2+ve invasive breast cancer that will not receive Herceptin
9. Bilateral invasive malignancy of the breast (synchronous or metachronous)
10. More than one primary tumor in different quadrants of the same breast
11. Presence of an ipsilateral breast implant or pacemaker
12. Status for adjuvant systemic therapy not determined
13. Unable to commence radiation therapy:

    1. within 12 weeks of the last surgical procedure on the breast, or
    2. within 8 weeks of the last dose of chemotherapy
14. Previous or concurrent malignancies except:

    1. Non-melanoma skin cancer
    2. Carcinoma in-situ of the cervix
    3. Invasive carcinoma of the cervix, endometrium, colon and thyroid, treated 5 years prior to study entry with no evidence of disease
15. Serious non-malignant disease (e.g. cardiovascular, pulmonary, systemic lupus erythematosus (SLE), scleroderma) which would preclude definitive radiation treatment.
16. Current pregnancy or lactating.
17. Psychiatric or addictive disorders which would preclude obtaining informed consent or adherence to the protocol.
18. Geographic inaccessibility for follow-up.
19. Inability to localize surgical cavity on CT (i.e. no evidence of surgical clips or seroma)
20. Inability to adequately plan the patient for the experimental technique.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Adverse cosmetic outcome using the EORTC Breast Cosmetic Rating System | 2 years post randomization
  The primary outcome is adverse cosmesis assessed at 2 years post randomization as determined by photographic assessment. The cosmetic outcome will be assessed by a panel of 3 trained radiation oncologists who are unaware of treatment allocation, using the EORTC Breast Cosmetic Rating System for cosmetic results for breast conserving treatment. The treated breast is compared with the untreated breast for size, shape, location of the areola/nipple, appearance of the surgical scar, presence of telangiectasia, and a global cosmetic score based on these factors. Characteristics are graded on a 4-point scale: 0 = excellent; 1 = good; 2 = fair; 3 = poor. A global cosmetic score of fair or poor will be used as the primary outcome of adverse cosmesis.

SECONDARY OUTCOMES:
Cosmetic deterioration (defined as any adverse change in the global cosmetic score) | Baseline to two years
  defined as any adverse change in the global cosmetic score from baseline to 2 years. Subjects with global cosmetic scores that were stable or improved from baseline to 2 years will be scored as 'no deterioration'.
Radiation toxicity assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v.4.02 | 12, 24, 36 and 60 months
  defined as breast induration/fibrosis, shrinkage, and telangiectasia, which will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v.4.02.
Ipsilateral breast tumour recurrence (IBTR) | Ongoing throughout study up to 5 years
  defined as recurrent invasive or in situ cancer in the ipsilateral breast including the axillary tail. Histological evidence of local recurrence will be required.
Disease free survival (DFS) | Ongoing throughout study up to 5 years
  defined as the time from randomization to the time of documented recurrent disease in the ipsilateral breast or regional nodes (supraclavicular, axillary or internal mammary) or distant sites (e.g. bone, liver, lung or brain).
Overall survival (OS) | From date of randomization until the date of death up to 5 years
  defined as the time from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Do-Hoon Kim, MD, Principal Investigator — Juravinski Cancer Centre
Locations (10):
- Canada (10):
  - Simcoe Muskoka Regional Cancer Centre, Royal Victoria Hospital, Barrie, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Regional Cancer Program; London Health Sciences Centre, London, Ontario
  - Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - CHUM Centre Hospitalier de L'Université de Montréal, Montreal, Quebec
  - CHUQ Pavillon Hotel-Dieu Quebec, Québec, Quebec
  - CHUS - Hopital Fleurimont, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim DH, Theberge V, Parpia S, Kong I, Provencher S, Yassa M, Perera F, Lavertu S, Rousseau P, Lee J, Karam I, Schneider K, Levine MN, Whelan TJ; OPAR Study Investigators. OPAR: A Randomized Trial of Partial Breast Irradiation in Five Fractions Once Daily for Early Breast Cancer. J Clin Oncol. 2025 Feb 10;43(5):505-512. doi: 10.1200/JCO.24.00600. Epub 2024 Oct 8. PMID 39378393